CLINICAL TRIAL: NCT00947466
Title: A Multi Centre Open Label Single Therapy Dose Ranging Study to Characterise the Pharmacokinetics & Tolerability of BTDS 5-20 ug/h in Children Who Require Opioid Analgesia for Moderate to Severe Mouth Pain Secondary to Chemotherapy Induced Mucositis.
Brief Title: A Study to Characterize the Pharmacokinetics and Tolerability of Buprenorphine Patches in Children With Moderate to Severe Mouth Pain
Acronym: BUP1501
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: 25 patients have been recruited and it was considered that further recruitment would add no extra PK information
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUP1501; 2008-002428-27
Record Dates: First submitted 2009-07-08; First posted 2009-07-28 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Chemotherapy Induced Mucositis; Mouth Pain
Keywords: Buprenorphine transdermal patch (BTDS); Moderate to severe mouth pain; Chemotherapy induced mucositis; Pharmacokinetic
MeSH Terms: interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patch (Experimental)
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — Transdermal patch

SUMMARY:
The purpose of this study is to characterize the pharmacokinetics and tolerability of buprenorphine patches in children who require opioid pain relief for moderate to severe mouth pain.

DETAILED DESCRIPTION:
Subjects will be screened for eligibility and if eligible will apply a buprenorphine patch (Day 1). The patch will be worn for 7 days during which time, safety assessments, pain scores, mucositis scores, PK sampling & vital signs will be assessed on each day. After patch removal subjects will continue with these assessments on a daily basis until Day 12. The subject will then be followed up for 10 days (to Day 22) to collect information on ongoing/new SAEs/AEs.

ELIGIBILITY:
Inclusion criteria:

1. Male or female children experiencing severe mouth pain secondary to chemotherapy induced mucositis requiring opioid analgesic therapy and who will be an inpatient, as a minimum up to Day 8 (patch removal).
2. Subjects experiencing 'severe' pain in the Investigators clinical judgment.
3. Body weight ≥ 15 kg. Subjects weighing ≥ 25 kg will be recruited in the first phase of the study with those weighing < 25 kg also being included in the second phase, (after a successful review by an IDSMC). Upper age range to be 16 years.
4. In dwelling IV cannula or central line from which blood can be obtained.
5. Written informed consent obtained from parent(s)/legal representative, and where possible assent obtained from the subject if appropriate, in line with local regulations.
6. Females of child bearing potential must have a negative urine pregnancy test if the Principal Investigator considers there to be a reasonable possibility of pregnancy.

Exclusion criteria:

1. Subjects with known hypersensitivity to buprenorphine or any of its excipients in the transdermal system, as outlined in the Summary of Product Characteristics for BuTrans.
2. Known hypersensitivity to other opioids.
3. Skin disease affecting application or local tolerance of BTDS.
4. Clinically significant history of allergic reaction to wound dressings or adhesives.
5. Severe respiratory impairment.
6. Clinically significant hepatic dysfunction.
7. Severe renal impairment.
8. Subjects who are receiving MAO inhibitors or have taken them within the previous 2 weeks.
9. Subjects receiving hypnotics or other central nervous system (CNS) depressants that, in the investigator's opinion, may pose a risk of additional CNS depression with study medication.
10. Subjects who have taken any buprenorphine preparations in the last 14 days.
11. Subjects with myasthenia gravis.
12. Subjects with convulsive disorders, head injury, shock, or reduced level of consciousness of uncertain origin.
13. Subjects who are currently participating in another clinical research study involving a new chemical entity (NCE) unless the sole purpose of the other trial at the time of BUP1501 screening is for long term follow-up/survival data or subjects who have participated in a clinical study within the previous 30 days. Participation in a chemotherapy clinical trial that is not evaluating a NCE will be accepted for inclusion.
14. Subjects who are pregnant, lactating or in the Investigators opinion are at risk of conceiving.
15. Previous enrollment in this clinical study.
16. Subjects who the Investigator believes are unsuitable for the study.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2010-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
To characterise the pharmacokinetics of BTDS 5-20 ug/h in children weighing >15kg | PK's taken daily for 12 days

SECONDARY OUTCOMES:
safety & tolerability of BTDS 5-20ug/h in children | every 4 hours to day 5, day 12 and day 21

CONTACTS AND LOCATIONS:
Locations (2):
- Skejby, Denmark
- Dr Howell, Liverpool, United Kingdom

REFERENCES:
- See also: Results available onw ebsite — https://www.clinicaltrialsregister.eu/ctr-search/search?query=BUP1501